CLINICAL TRIAL: NCT04696835
Title: Use of Near-infrared Functional Spectroscopy (fNIRS) in the Evaluation of Hearing Rehabilitation in Children With Hearing Aid(s)
Brief Title: fNIRS in Pediatric Hearing Aids
Acronym: FNIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Fondation William Demant (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018_73; 2019-A02517-50 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss
Keywords: NIRS; hearing aid; pediatrics; cochlear implant; rehabilitation; neuroimaging
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry, Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children with hearing aids (Experimental)
  Interventions: Diagnostic Test: speech audiometry
- control group (Sham Comparator)
  Interventions: Diagnostic Test: speech audiometry

INTERVENTIONS:
Diagnostic Test: speech audiometry — 65dB, 55dB or 75dB SPL speech audiometry

SUMMARY:
Pilot phase. Monocentric, non-controlled, non-randomized, open-label study evaluating the capacity of the functional near-infrared functional neuroimaging (fNIRS) technique to translate temporal cortical activity in response to a speech stimulus in normo-hearing and deaf children with cochlear implants.

Hemodynamic changes are expected to be observed that indicate brain activity following the stimuli, resulting in a change in the concentration of oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) recorded by the fNIRS.

The use of the FNIRS in the evaluation of hearing aid effectiveness could contribute to a more adapted management of childhood hearing loss since conventional methods in young children are not adapted to the needs of children with hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Infants and toddlers 3-18 months of age who are normal hearing.
* Group B: Infants and toddlers aged 3 to 18 months with sensorineural hearing loss fitted with a unilateral or bilateral hearing aid with optimized adjustments by the hearing healthcare professional.
* Socially insured subject
* Parents or guardians who have given their consent to participate in the study

Exclusion Criteria:

* Medical condition that does not allow for research compliance.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Oxygenated haemoglobin concentration (HbO) | Baseline (at inclusion)

SECONDARY OUTCOMES:
Deoxygenated haemoglobin concentration (HbR) | Baseline (at inclusion)
HbO Concentration | At 3 months, 6 months, 12 months and 24 months
  Evolution of the variation in HbO concentration in the group of infants fitted with a device.
HbR Concentration | At 3 months, 6 months, 12 months and 24 months
  Evolution of the variation in HbR concentration in the group of infants fitted with a device.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe VINCENT, PU-PH, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France